CLINICAL TRIAL: NCT05799001
Title: Dance Workshop for Institutionalized Seniors With Behavioral and Psychological Symptoms of Dementia
Acronym: APAISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Emile Roux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RIPH2_CHAPPUIS_APAISE; 2022-A02335-38 (Other: ID-RCB)
Record Dates: First submitted 2023-03-03; First posted 2023-04-05 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — Dance Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): 4 months of dance workshop with a Professional dance teacher
  Interventions: Behavioral: Dance therapy
- Control (Other): First, patients will have usual activities for 4 months and in a second time, they will have 4 months of dance class with a nurse previously trained by the dance teacher
  Interventions: Behavioral: Dance therapy

INTERVENTIONS:
Behavioral: Dance therapy — Patients will be randomized in 2 groups, experimental or control.
  The experimental group will have 4 months of dance therapy with a professional dancer and will then resume there usual activities.
  The control group will start with their usual activities in the nursing home for the first 4 months and then, they will have dance sessions with a nurse previously trained by the dancer.

SUMMARY:
It is estimated that the prevalence of dementia in France is 5% for people over 65 years of age and that this increases to 18% for people over 75 years of age. Behavioral disorders are frequent in patients with dementia and are the main cause of institutionalization, representing up to 50% of cases. Dementia syndromes can be translated into behavioral and psychological symptoms of dementia (BPSD), which are defined as perceptual, mood or behavioral disorders. To date, there is no cure for dementia, but certain measures can be taken to reduce symptoms. The HAS suggests that physical exercise would reduce BPSD and could improve the ability to perform activities of daily living or slow down the cognitive decline of this type of patient. Indeed, several articles have highlighted the benefits of physical activity in demented patients. A meta-analysis has shown a significant decrease in BPSD via the Neuropsychiatric Inventory (NPI) score. Nevertheless, it is often observed that there is a difficulty in adhering to the program in very elderly population groups. Dance is a complete physical activity that integrates physical, cognitive and social elements. A meta-analysis has shown that dance has a significant effect on global cognition but also on neuroplasticity and physical functioning in patients with mental disorders. The music component of dance also has an effect on the behavioral problems of demented patients, stimulating language ability and social and emotional function.

However, at present, no study of good methodological quality has been able to demonstrate the effectiveness of dance-based physical activity for the treatment of dementia symptoms. As a result of these findings, the APAISE project was developed and should help slow the onset of BPSD in patients with dementia.

ELIGIBILITY:
Inclusion Criteria:

1. Institutionalized patient (male or female) over 65 years of age ;
2. Patient with behavioral problems, as measured by an NPI-ES ≥ 4 on any item and an NPI-ES impact scale ≥ 3 ;
3. Patient able to mobilize the upper body at a minimum (arms, trunk, head);
4. Medication (antipsychotics, antidepressants, anxiolytics and related hypnotics) without major modification for at least 30 days prior to inclusion after medical advice;
5. Possibility of including patients under guardianship or curatorship;
6. Patient affiliated to a social security plan;
7. Obtaining consent from the patient or legal representative.

   Exclusion Criteria:
8. Inability of the patient to follow the sessions (e.g., major visual/auditory disabilities), difficult follow-up, or any other reason at the discretion of the investigator;
9. Inability of the health care team to complete the NPI-ES questionnaire for the patient;
10. Patient has a concurrent psychiatric disorder (e.g., bipolar disorder, schizophrenia, or other).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Compare the effectiveness of adding biweekly dance class for 4 months on behavioral and psychological symptoms of dementia in institutionalized older adults compared to usual care alone. | 4 months
  The primary endpoint was the overall score on the validated Neuropsychiatric Inventory questionnaire, completed by the health care teams. This questionnaire will be done at inclusion (day 0) and after 4 months of dance therapy for the experimental group or usual care alone for the control group.This questionnaire allows to highlight behavioral disorders in patients suffering from dementia according to 10 behavioral domains and 2 neurovegetative variables (sleep and appetite).

SECONDARY OUTCOMES:
evolution of behavioral problems | - 8 and 12 months for the experimental group- 12 and 16 months for the control group
  Neuropsychiatric Inventory (NPI-ES) score
evaluation of cognitive functions | - 4 months (for the 2 groups)- 8 and 12 months for the experimental group- 12 and 16 months for the control group
  Mini Mental State Examination (MMSE) score. The questionnaire consists of 30 items, and each correct answer is worth 1 point. The score must take into account the patient's age and level of education.
autonomy or degree of dependence | - 4 months (for the 2 groups)- 8 and 12 months for the experimental group- 12 and 16 months for the control group
  Activities of Daily Living (ADL) score. This questionnaire studies the autonomy or degree of dependence of institutionalized patients in carrying out practical activities of daily living: personal hygiene, dressing, going to the toilet, locomotion, continence, eating. It is made up of 6 items, and each item has 3 possible answers. Answers must correspond to the patient's abilities. A total score of 6 indicates maximum patient autonomy.
activity frequency of dementia patients | - 4 months (for the 2 groups)- 8 and 12 months for the experimental group- 12 and 16 months for the control group
  Activity and Affect Indicators of Quality of Life (AAIQOL) score This questionnaire contains 21 items: 15 items relating to patient activity and 6 items relating to patient affect. The questionnaire highlights decreases in the frequency of activity in institutionalized dementia patients, as well as increases in negative affect and decreases in positive affect, both of which are indicators of worsening dementia.
state of depression | - 4 months (for the 2 groups)- 8 and 12 months for the experimental group- 12 and 16 months for the control group
  short-Geriatric Depression Scale (short-GDS) score This questionnaire is used to assess depression in the elderly and demented. The short-GDS is a shortened version (15 items) of the GDS (30 items). Each item is answered with a yes or no. Depending on the answer, a value of 0 or 1 is assigned. A total score between 0 and 5 is considered normal, between 5 and 9 indicates probable depression, and a score greater than or equal to 10 almost always indicates the existence of depression.
minimal motor and postural possibilities | - 4 months (for the 2 groups)- 8 and 12 months for the experimental group- 12 and 16 months for the control group
  Test Moteur Minimum (TMM) score This simple clinical test can be used to assess the minimum motor and postural capabilities of frail elderly subjects. The test assesses postural skills and protective reactions of the upper and lower limbs. Scoring calls for an affirmative or negative response. Each response is assigned a score: if the response is in favor of preserved motor capacity, the score is 1, whereas the score is 0 if the response is in favor of abnormal motor aptitude. This results in an overall score out of 20. The 20 items are divided into 4 themes: - decubitus mobility; - sitting; - standing; - walking. Retropulsion is demonstrated in this test in the sitting, standing and walking positions.
collection of drugs | - 4 months (for the 2 groups)- 8 and 12 months for the experimental group- 12 and 16 months for the control group
  collected on the medical record : antipsychotics, antidepressants, anxiolytics and related hypnotics
program membership | 12 months for the experimental group16 months for the control group
  Refusal rate for participation in dance workshops
program membership | 12 months for the experimental group16 months for the control group
  Rate of premature discharge or lost sight
program membership | 12 months for the experimental group16 months for the control group
  Number of sessions attended by patients.
contribution of dance-based physical activity for trained caregivers | 8, 12 and 16 months
  evaluated by :
  - A satisfaction questionnaire
contribution of dance-based physical activity for trained caregivers | 8, 12 and 16 months
  evaluated by :
  - Semi-structured interviews
contribution of dance-based physical activity for trained caregivers | 8, 12 and 16 months
  evaluated by :
  - Number of sessions realised independently
contribution of dance-based physical activity for trained caregivers | 8, 12 and 16 months
  evaluated by :
  - Number of patients attending sessions
contribution of dance-based physical activity for trained caregivers | 8, 12 and 16 months
  evaluated by :
  - Frequency of sessions realised.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Pays Craponne, Craponne-sur-Arzon
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay